CLINICAL TRIAL: NCT07004283
Title: Fetal Magnetic Resonance Imaging: Z-score Reference Ranges for a Large Patient Population in Normal Neuroimaging Measurement
Acronym: FMZSCORE
Status: Enrolling by invitation | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025282B00
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Fetal Growth Retardation; Fetal Neurodevelopmental Disorder
Keywords: z-score; healthy reference range
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to establish the z score reference ranges of fetal head circumference and other measurement of fetal measurements including biparietal diameter, fronto-occipital diameter, length of the corpus callosum, lateral ventricle, transverse cerebellar diameter, height of the vermis, anteroposterior diameter of the vermis，height and width of normal fetuses from 18 to 40 weeks' gestation.

Method-A cohort-based study was conducted on low-risk singleton pregnancies with healthy fetuses. The measurement was performed using simple 2-dimensional MRI on the typical fetal standard view. The reference ranges were constructed according to gestational age (GA), biparietal diameter (BPD), as independent variables based on the best-fit models, both mean and standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

* The pregnant women in Born in Guangzhou Cohort Study

Exclusion Criteria:

* The fetuses with prenatal diagnosis of congenital heart disease or other congenital diseases.

The fetuses who are high-risk neonates at the delivery.1) preterm infants; (2) infants with extremely low birth weight (ELBW) or who are small for gestational age (SGA);

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was based on the Born in Guangzhou Cohort Study (BIGCS), a prospective cohort study conducted in Guangzhou, China. The protocol of BIGCS was described in detail previously [20]. In brief, women who planned to give birth at the Guangzhou Women and Children's Medical Center and live in Guangzhou for at least 3 years after delivery were invited to participate in the BIGCS at their first antenatal visit (< 20 weeks' gestation). The study was approved by the Institutional Ethics Committee of the Guangzhou Women and Children's Medical Center. Before recruitment, written informed consent was obtained from all participants.
  Inclusion criteria for the current study were (1) pregnant women aged 18 years or above, (2) singleton pregnancies and (3) pre-pregnancy BMI < 18.5 kg/m2. The exclusion criteria were as follows: (1) withdrew before delivery, (2) diagnosed with diabetes, hypertension, and heart disease before pregnancy, (3) terminations of pregnancy or stillbirths, (4) multiple g
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Birth | 20 weeks follow up
  Healthy birth

SECONDARY OUTCOMES:
low birth weight | 20 weeks follow up
  Healthy birth

CONTACTS AND LOCATIONS:
Locations (1):
- Siemens Skyra 3.0T MRI, Guangzhou, Guangdong, China